CLINICAL TRIAL: NCT01690741
Title: A Phase 1, Open-Label, Dose-Escalation Study Evaluating the Safety, Pharmacokinetics, Pharmacodynamics, and Clinical Effects of Intravenously Administered Nerofe™ in Subjects With Advanced Malignancies
Brief Title: Phase 1 Trial of Intravenously Administered Nerofe™ in Subjects With Advanced Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Immune System Key Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ISK-N101
Record Dates: First submitted 2012-09-12; First posted 2012-09-24 (Estimated); Last update posted 2018-06-25 (Actual); Status verified 2018-06

CONDITIONS: Cancer
Keywords: Cancer; Malignancy; Solid tumors
MeSH Terms: conditions — Neoplasms | interventions — tumor-cells apoptosis factor, human

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Nerofe (Experimental): Nerofe administered intravenously 3x/week
  Interventions: Drug: Nerofe

INTERVENTIONS:
Drug: Nerofe — Nerofe administered intravenously 3x/week
  Other Names: Tumor-Cells Apoptosis Factor

SUMMARY:
This study will be the first to test the anti-cancer peptide Nerofe in humans. It will evaluate the safety, pharmacokinetic behavior, and pharmacodynamic and clinical effects of Nerofe given intravenously every other day to patients with advanced malignant disease.

DETAILED DESCRIPTION:
This is a Phase 1 single-center, open-label, non-randomized, dose-escalation study, to be conducted in 2 phases. The Dose Escalation Phase will determine the maximum tolerated dose (MTD) of Nerofe and evaluate its safety and tolerability, pharmacokinetics, pharmacodynamics, immunogenicity, and preliminary clinical effects. The subsequent Dose Confirmation Phase will be a cohort expansion at or below the MTD of Nerofe. Subjects will be treated with IV doses of Nerofe thrice weekly (on alternating days) in consecutive, 28-day cycles. Subjects will be evaluated regularly for safety. Subjects who tolerate the drug and who do not experience progressive disease, intolerable toxicity, or meet any of the other withdrawal criteria may continue to receive Nerofe for up to 6 cycles, at the discretion of the Principal Investigator. Throughout the trial, oversight will be provided by the Clinical Safety Committee.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all of the following inclusion criteria to be eligible for the study:

1. Males and females above 18 years of age.
2. Pathologically confirmed locally advanced and/or metastatic solid tumor for which, in the judgment of the Principal Investigator, no standard curative therapy exists.
3. Beginning with Cohort 6 of the Dose Escalation Phase and beyond, including the Dose Confirmation Phase, subjects must have 1 of the following solid tumor types: renal cell carcinoma, ovarian carcinoma, triple-negative breast cancer, or metastatic colorectal carcinoma.
4. Disease that is evaluable measurable on physical examination or imaging by Response Evaluation Criteria in Solid Tumors (RECIST v1.1 Appendix A), or is characterized by informative tumor marker(s).
5. Eastern Cooperative Oncology Group (ECOG) Performance Status ≤ 1 (Section 9.1.1.6).
6. Acceptable clinical laboratory values at screening, as indicated by:

   * Absolute neutrophil count ≥ 1,500/mm3;
   * Platelets ≥ 75,000/mm3;
   * Total bilirubin ≤ 1.5 × the upper limit of normal (ULN);
   * AST (SGOT) ≤ 2.5 × the ULN;
   * ALT (SGPT) ≤ 2.5 × the ULN;
   * Serum creatinine ≤ 1.5 mg/dL or a measured creatinine clearance ≥ 60 mL/min; and
   * Negative serum Beta hCG test in women of childbearing potential (defined as women ≤ 50 years of age or history of amenorrhea for ≤ 12 months prior to study entry).
7. Patients with hepatic metastasis are eligible to enroll, provided that the following criteria are met at Screening:

   * Total bilirubin is no higher than the ULN;
   * AST and ALT are each ≤ 5 × the ULN;
   * Severe liver dysfunction (Child-Pugh Class B or C) is not present; and
   * Patients with a history of esophageal bleeding have varices that have been sclerosed or banded and no bleeding episodes have occurred during the prior 6 months.
8. If there is a history of brain metastasis treated with radiation therapy, the radiation therapy must have been completed at least 4 weeks prior to enrollment, the metastatic disease must have been stable since completion, and the subject maybe taking no more than 4 mg/day of dexamethasone
9. Willing and able to provide written Informed Consent and comply with the requirements of the study.
10. Beginning with Cohort 5 of the Dose Escalation Phase: Tumor tissue, taken from either an archival sample or a fresh biopsy, must be available for staining for T1/ST2 receptor (see Sections 8.2.1 and 8.2.3).
11. In the Dose Confirmation Phase only, subjects must have disease that is measurable on physical examination or imaging by RECIST v1.1 (Appendix A).

Exclusion Criteria:

1. Any chemotherapy, immunomodulatory drug therapy, anti-neoplastic hormonal therapy (unless dose has been stable for 3 months prior to Baseline and remains stable during the trial), immunosuppressive therapy, corticosteroids > 20 mg/day prednisone or equivalent (unless administered to prevent contrast material reactions during radiographic procedures), or growth factor treatment (eg, erythropoietin) within 14 days prior to initiation of study drug.
2. Presence of an acute toxicity of prior chemotherapy, with the exception of alopecia or peripheral neuropathy, that has not resolved to ≤ Grade 1, as determined by NCI CTCAE v 4.0 (http://evs.nci.nih.gov/ftp1/CTCAE/About.html).
3. Receipt of >2 prior regimens of cytotoxic chemotherapy, including any use in the neo-adjuvant, adjuvant, and/or metastatic settings.
4. Life expectancy <12 weeks.
5. Major surgery or radiation therapy within 28 days prior to initiation of study drug, or highly localized radiation therapy for symptoms control within 14 days of initiation of study drug.
6. Receipt of radiotherapy to >25 % of bone marrow.
7. Known human immunodeficiency virus (HIV) or acquired immunodeficiency syndrome-related illness.
8. Known active hepatitis B or C or other active liver disease (other than malignancy).
9. Active infection requiring systemic therapy.
10. Insulin-requiring diabetes mellitus.
11. History of any of the following within 12 months prior to initiation of study drug:

    Uncontrolled congestive heart failure (New York Heart Association Classification 3 or 4), unstable angina, myocardial infarction, cerebrovascular accident, coronary/peripheral artery bypass graft surgery, transient ischemic attack, or pulmonary embolism.
12. Uncontrolled arterial hypertension, or anti-hypertensive drugs whose type or dose has been changed within 3 months prior to screening or whose dose is anticipated to change within cycle 1.
13. History of syncope, pre-syncope or orthostasis.
14. Risk of syncope, in the judgment of the Principal Investigator.
15. History of or ongoing cardiac dysrhythmias requiring treatment, atrial fibrillation of any grade, or persistent prolongation of the QTc (Fridericia) interval to > 450 msec for males or > 470 msec for females.
16. Previous malignancy, except for intraepithelial neoplasia; basal cell carcinoma of the skin; adequately treated localized prostate carcinoma with current Prostate-Specific Antigen <1.0 ng/mL; a history of potentially curative therapy with no evidence recurrence for at least 2 years; or a previously treated malignancy within the past 2 years that the Principal Investigator deems to be at low risk for recurrence during the course of this trial.
17. Use of any investigational agents within a minimum of 3 weeks or 5 half-lives of initiation of study drug.
18. Pregnant or lactating female.
19. Women of childbearing potential, unless they agree to use dual contraceptive methods which, in the opinion of the Principal Investigator, are effective and adequate for that patient's circumstances while on study drug and for 3 months afterward.
20. Men who partner with a woman of childbearing potential, unless they agree to use effective, dual contraceptive methods (ie, a condom, with female partner using oral, injectable, or barrier method) while on study drug and for 3 months afterward.
21. Any severe, acute, or chronic medical or psychiatric condition, or laboratory abnormality that may increase the risk associated with study participation or study drug administration, may interfere with the informed consent process and/or with compliance with the requirements of the study, or may interfere with the interpretation of study results and, in the investigator's opinion, would make the patient inappropriate for entry into this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2013-12 (Actual); Primary Completion 2017-12-19 (Actual); Study Completion 2017-12-19 (Actual)

PRIMARY OUTCOMES:
Safety, as determined by frequency, nature, and severity of adverse events; and the profile of dose-limiting toxicities | Up to 6 months

SECONDARY OUTCOMES:
Pharmacodynamic effects of Nerofe, through the measurement of serum concentrations of biomarkers (including cytokines and circulating soluble T1/ST2 receptor) and peripheral blood mononuclear cell expression of T1/ST2 receptor | Up to 6 months
Clinical effects of Nerofe on cancer, as assessed by Response Evaluation Criteria in Solid Tumors | Up to 6 months
Pharmacokinetic behavior of Nerofe: plasma concentrations in ng/mL | Pre-dose (Cycle 1 Days 1 and 29 only); and 0.25, 1, 2, 4h, 6, 8, and 24h following the end of infusion (Cycle 1 Days 1 and 29)
Pharmacokinetic behavior of Nerofe: plasma half-life in minutes | Cycle 1 Day 1 and Day 29
Relationship between pretreatment fresh/archival tumor tissue T1/ST2 receptor expression and biological activity of Nerofe | Up to 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Yoram Devary, PhD, Study Director — Immune System Key Ltd
Locations (1):
- Kaplan Medical Center, Rehovot, Israel

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Sandler U, Devary O, Braitbard O, Ohana J, Kass G, Rubinstein AM, Friedman ZY, Devary Y. NEROFE--a novel human hormone-peptide with anti-cancer activity. J Exp Ther Oncol. 2010;8(4):327-39. PMID 21222365
- See also: Immune System Key Ltd. Website — http://www.immunesk.com/